CLINICAL TRIAL: NCT06437080
Title: Hypoferritinemia Without Anemia Among Reproductive Age Females: Frequency, Determinants and Treatment Outcomes
Brief Title: Hypoferritinemia Without Anemia Among Reproductive Age Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akram Medical Complex (Other)
Collaborators: Scotmann Pharmaceuticals (Industry); The Searle Company Limited Pakistan (Industry)
Responsible Party: Principal Investigator, Shehla Javed Akram, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70122031
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hypoferritenemia Without Anemia (HWA); Iron Deficiency Without Anemia)
Keywords: Hypoferritenemia without Anemia (HWA); Reproductive age females; Symptoms of HWA; Determinants of HWA; Low serum ferritin levels, Iron deficiency; Cross-sectional study (Phase 1); Randomized controlled trial (Phase 2); Transferrin saturation (TSAT); Intervention
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: After randomization, 100 patients will be allocated to each of the three study groups, (total participants selected 300) i.e., group A, B and C.
  The participants of Group A will get oral Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron, 100 mg (Fersip) daily for three months, participants of group B will get IV Ferric Carboxymaltose (Ferinject) for 03 months (3 doses) and Group C will remain on their normal diet
  All 03 groups will be called and their blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and severity of symptoms to assess the effectiveness of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral iron supplement (Active Comparator): 100 participants of Group A will get oral iron supplementation (Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron), 100 mg for 03 months. Participants will consume 01 tablet per day for 03 months.
  After completion of the treatment period blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and severity of symptoms to assess the effectiveness of the intervention.
  Interventions: Drug: Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron, 100 mg
- Intravenous (IV) iron supplementation (Active Comparator): 100 participants of Group B will get IV iron supplementation (Ferric Carboxymaltose) for 03 months (01 dose per month for 03 months).
  After completion of the treatment period blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and severity of symptoms to assess the effectiveness of the intervention.
  Interventions: Drug: Ferric Carboxymaltose
- Normal diet (No Intervention): 100 participants will remain on their normal diet for 03 months. After 03 months blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and severity of symptoms to assess the effectiveness of the intervention.

INTERVENTIONS:
Drug: Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron, 100 mg — 01 tablet daily for 03 months, This is assigned to Group A.
  Other Names: Fersip
  Arms: Oral iron supplement
Drug: Ferric Carboxymaltose — 03 doses (50 mg iron/mL) per month for 03 months. This is assigned to Group B.
  Other Names: Ferinject
  Arms: Intravenous (IV) iron supplementation

SUMMARY:
The goal of this randomized controlled trial is to compare the treatment outcomes of oral iron supplementation (Group A) versus Intravenous (IV) iron supplementation (Group B) versus normal diet (no treatment) (Group C) on the serum ferritin level and to determine the outcomes in the severity of symptoms of HWA, among reproductive age females (age 18-45) with hypoferritinemia without Anemia (HWA), after four months of the start of the intervention.

The main questions it aims to answer are:

1. What are the main determinants of HWA?
2. There is no difference/ difference in the treatment outcomes after intervention
3. There is no difference/ difference in the severity of symptoms of HWA after intervention.

Participants will:

* Randomly divided into 3 groups (A, B and C) to receive treatment.
* 100 patients will be allocated to each of the three study groups i.e., group A, B and C. The participants of Group A will get oral Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron, 100 mg (Fersip) daily for three months, participants of group B will get IV Ferric Carboxymaltose (Ferinject) for 03 months (3 doses) and Group C will remain on their normal diet,
* Visit the clinic once every 1 month for 03 months for doses and assessment of symptoms and adverse events will be done.
* All 03 groups will be called after one month of the last dose and the blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and the severity of symptoms to assess the effectiveness of the intervention.

DETAILED DESCRIPTION:
At present the commonly identified presentation is Iron Deficiency Anemia which currently affects more than 1 billion people while Hypoferritenemia without Anemia (HWA) is at least twice as common. HWA is poorly recognized by clinicians despite its high prevalence, probably because of suboptimal screening recommendations.

HWA: Patients having normal Hemoglobin of ≥12 g/dl and having below normal range ferritin level < 30ng/ml and patients suffering from any of the following symptoms of

* Fatigue/ tiredness
* Poor work productivity
* Poor attention
* Poor memory
* Sore tongue
* Poor condition of skin, nails or hair, including hair loss.
* Delayed skin wound healing
* Palpitation
* Restless Leg Syndrome

As the symptoms and signs of the HWA are nonspecific which may happen in other systemic diseases or psychiatric disorders so patients with HWA are either recommended no tests or later on end up with expensive tests for heart failure and renal failure on the other end which can be the result of chronic iron deficiency. Clinicians usually advise iron studies when there is documented anemia which results in underdiagnoses of HWA.

In United Kingdom, National Diet and Nutrition Survey (2008/2009-2011/2012) were conducted. The study found that around 15·5 % of women of 19 to 64 years of age had serum ferritin levels < 15ng/ ml (Adams & White, 2015). Another National survey conducted in US found that around 11% of the women belonging to 18 to 49 years of age had plasma ferritin levels < 12ng/ ml.

In another study conducted in Iran 2020, serum ferritin levels were observed among 120 females. The sample was selected from the outpatient department of a medicine clinic. The blood samples of the participants were obtained to have a complete account of their CBC and serum ferritin levels. Results revealed that 41.7% of the patients had severe iron deficiency with low level of serum ferritin values (value <10ng/ml). Among symptoms of iron deficiency, the most common symptom reported among 79.2% patients was fatigue. Other symptoms include hair loss reported by 73.3%, dizziness reported by 70.0%, headache reported by 65.8%, poor concentration reported by (61.7%), palpitation by (60.0%), chest pain by (55.8%) and legs pain by (47.5%) of the participants. Among females of younger age group (less than 25 years), lower levels of serum ferritin were associated with heavy menstrual bleeding. Whereas, among females of older age group (above 25 years of age) poor nutrition reported to be a significant risk factor of low serum ferritin values. In conclusion, the study addressed low serum ferritin without anemia as a concealed disease that should be addressed by considering its treatment and diagnosis because patients with normal hemoglobin levels can develop iron deficiency anemia within days after diagnosis.

To the best of researcher's knowledge, no study related to HWA has been conducted in Pakistan; therefore, the prevalence of Iron Deficiency Anemia (IDA) in Pakistan has been added in the present literature review. Results show that a total of 45% of population is suffering from IDA in Pakistan.

The rationale of this study is to highlight the struggling issue of HWA which is battling to be recognized as one of the factors contributing to the symptoms indicated above, as was previously stated. This study is important to be conducted as it will not only pave ways to recognize the category of HWA but will also help patients to receive targeted treatment and saving them from the risk of drug abuse and over-medication. As per the researcher's knowledge, there is a scarcity of data on Pakistan's population as no study exists on HWA in Pakistan.

Above literature review clearly reflects that there is a wide gap regarding some aspects of HWA. First, it is an underdiagnosed entity as it has nonspecific symptoms which can be found in other diseases. Although there are estimates of disease burden, but exact value is not known especially in developing countries. Secondly, there is a lot of data regarding causes of iron deficiency but paucity exists regarding determinants/causes of HWA. Thirdly, there is contrary data regarding management, few investigators believe that oral iron therapy shall be the first line therapy while other believes that intravenous (IV) therapy shall be given first to reduce symptoms.

OBJECTIVES

1. To determine the frequency and Determinants of HWA among women of reproductive age
2. To compare the treatment outcomes of oral iron supplementation (Group 1) versus Intravenous (IV) iron supplementation (Group 2) versus normal diet (Group 3) on the serum ferritin level after four months of start of intervention
3. To determine the outcomes in the severity of symptoms of HWA after four months of start of intervention

DETERMINANTS OF HWA

* Heavy menstrual bleeding
* Blood donation history
* Blood transfusion history
* Dietary intake
* Number of pregnancies
* Current status of lactation
* Family history of Anemia
* History of blood diseases
* Medication history of vitamins, minerals, or any other supplementation
* History of Drugs intake
* Disturbed Thyroid level and Blood Sugar levels
* Various co-morbidities or clinical conditions including, celiac disease, hemorrhoids, malignancies, hematuria, heart disease, renal failure, chronic gastric symptoms/ gastric ulcers, delayed wound healing and chronic liver disease
* The Symptom Severity Scale is a self-administered questionnaire that has been adapted from Spies-Derglo et al., to assess the severity of symptoms in patients.

DATA COLLECTION TOOL

For data collection, a structured close-ended questionnaire will be used. The developed questionnaire has six sections.

1. The first section consists of 5 qualifying question asking about age, premature menopause, blood transfusion history, supplementation history and history of any symptom of HWA (Defined above).
2. The second section will record the socio-demographic characteristics of the participants including, education, monthly family income, region of residence, religion, working status, marital status and the number of children and the utilization of antenatal care if ever pregnant.
3. The third section will be used to record the determinants leading to low serum ferritin levels including blood donation history, current lactation and pregnancy status, number of pregnancies, family history of Anemia, Menorrhagia; heavy menstrual bleeding, blood diseases, history of intake of medication other than supplements and vitamins, history of co-morbidities, and frequency of meals per day. The dietary score will also be measured using an individual DDS questionnaire. The score of DDS will be then recoded into different categories (≤ 3 as low, 4-5 as moderate, and ≥ 6 as high dietary diversity) according to the "Guidelines for measuring household and Individual Dietary Diversity".
4. The fourth section will record the serum ferritin, CBC, thyroid and blood sugar levels of the participants determined through lab tests. Participants having Vitamin B12 deficiency, Folic Acid deficiency, serum ferritin values >10ng/mL, disturbed thyroid and blood sugar levels, any chronic conditions will not be included in RCT.
5. Fifth section will inquire about the severity of clinical symptoms of participants at Visit 1 using a symptom severity scale to record baseline data.
6. The last section will be used to record the occurrence of adverse events followed by the administration of supplementation dosage to the participants of group A and B at visits 2, 3, 4, and 5, Serum ferritin value at visit 5 and the incidence and severity of clinical symptoms of HWA among patients at visit 5. Last question in section six will enquire about the subjective knowledge of participants regarding improvement in their symptoms before and after the intervention.

DATA COLLECTION PROCESS Cross-Sectional Study Study participants will be selected from four hospitals of Lahore through simple random sampling technique. Patients will be enrolled after meeting inclusion and exclusion criteria and filling of questionnaire during face to face interviews. At the end of each interview, the blood sample will be taken. Their blood will be tested for CBC and serum ferritin values at the end of the face to face interview. Informed written consent will be taken from each respondent before the start of the interview.

Randomized Control Trial (RCT)

* Females having normal CBC, hemoglobin level above 12mg/dl and serum ferritin level below 30 ng/ml and normal thyroid and blood sugar levels will be selected for the intervention.
* Females will be randomly assigned to three study groups.
* After randomization, 100 patients will be allocated to each of the three study groups i.e., group A, B and C. The participants of Group A will get oral Iron III Hydroxide Polymaltose Complex eq. to Elemental Iron, 100 mg (Fersip) daily for three months, participants of group B will get IV Ferric Carboxymaltose (Ferinject) for 03 months (3 doses) and Group C will remain on their normal diet,
* Assessment of symptoms and adverse event will be done
* All 03 groups will be called and their blood samples will be taken to evaluate the effect of iron supplementation on serum ferritin levels and severity of symptoms to assess the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age females: 18 to 45 years
* Clinical symptoms of iron deficiency which are fatigue/ tiredness, poor work productivity, poor attention and memory loss, sore tongue, poor condition of skin, nails or hair, including hair loss, delayed skin wound healing, palpitation and restless leg syndrome
* Normal CBC: hemoglobin level12mg/dl and above
* Serum ferritin levels: below 30 ng/ml
* Normal thyroid levels
* Normal blood sugar levels
* Willing and able to sign informed consent

Exclusion Criteria:

* Males
* Post-menopausal
* Premature menopause
* Anemic Females: hemoglobin levels i.e. less than 12 g/dl
* Serum ferritin level above 30 ng/ml.
* Disturbed thyroid levels
* Disturbed blood sugar levels
* Pregnant
* Lactating
* Blood donors
* Co-morbidities i.e., celiac disease, hemorrhoids, malignancies, hematuria, ulcers, heart failure, renal failure, chronic gastric symptoms/ gastric ulcers, chronic liver disease, disturbed thyroid levels and diabetes
* Any medication or supplement which may impact iron metabolism.
* History of iron or multivitamins supplementation in the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females of reproductive age
Enrollment: 1331 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Symptom severity scale | Week 1 (Baseline)
  Symptom severity score before intervention: This questionnaire contains eight questions with multiple-choice responses, with a score ranging from 0 point (not at all), 1 point (mild symptoms/ rarely), 2 points (moderate/ sometimes) and 3 points (severe/ frequently). The total symptom severity score will be calculated as the mean of the scores for the eight individual items and will be recorded at week 1
Determinants of Serum Ferritin value | Week 1 (Baseline)
  A questionnaire will be use to access the determinants. The questions included are blood donation history, vitamin supplementation drug, medication history, total preganacies, currently pregnant or lactating, heavy menstural bleeding, number of days of menstural bleeding and pads changed, frequency of stools per day, family history of anemia, frequency of meals per day and meal skipping
Socio demographic characteristics of participants | Week 1 (Baseline)
  The characteristics that will be surveyed at level of education, region, religion, income, marital status, number of children, antenatal care and working status
Dietary Diversity questionnaire | Week 1 (Baseline)
  For pattern of diet intake: History regarding daily meal frequency and skipping meals and 24 hour recall dietary of an individual will be surveyed: The score of all food groups will then be computed to get the final DDS. DDS of ≤3 will be considered low, 4-5 will be considered as moderate and ≥6 will be considered as a high DDS.
Serum ferritin levels | Week 1 (Baseline)
  Serum ferritin levels before intervention
Hemoglobin levels | week 1 (Baseline)
  Complete blood count (CBC)
Thyroid-stimulating hormone (TSH) | Week 2
  Thyroid functions
Random blood sugar | Week 2
  blood sugar levels

SECONDARY OUTCOMES:
Adverse events | Week 6, 10, 16
  Defined as participants self-reported adverse effects. Items that will be surveyed are nausea, vomiting, diarhhea, fever and others.
Symptom severity scale | Week 6, 10, 16
  Change in symptoms severity score after intervention: This questionnaire contains eight questions with multiple-choice responses, with a score ranging from 0 point (not at all), 1 point (mild symptoms/ rarely), 2 points (moderate/ sometimes) and 3 points (severe/ frequently). The total symptom severity score will be calculated as the mean of the scores for the eight individual items and will be recorded at week 6, 10, 16
Change in serum ferritin levels as result of oral intervention: Fersip | Week 16
  Change in serum ferritin levels as the result 90 tablets for 03 months (01 tablet everyday for 03 months)
Change in serum ferritin levels as result of intravenous (IV) iron intervention: Ferinject | Week 16
  Change in serum ferritin levels as the result of 03 doses (500 mg) per month for 03 months. The change will be measured through serum ferritin blood test results.
Comparison of treatment outcomes of groups (A, B and C) | Week 16
  Comparison of treatment outcomes of oral and IV iron supplementation and normal diet: The treatment outcomes will be measured through serum ferritin test as a comparison between 03 arms. Adverse events will also be compared. Items that will be surveyed for adverse events are are nausea, vomiting, diarrhea, fever and others

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Abdul Majeed Akhtar, MBBS, PhD, Study Chair — The univeristy of Lahore; Dr. Rubeena Zakir, MBBS, PhD, Study Director — University of Punjab
Locations (4):
- Pakistan (4):
  - Fatima Memorial Hospital, Lahore, Punjab Province
  - General Hospital Lahore, Lahore, Punjab Province
  - Gulab Devi Hospital, Lahore, Punjab Province
  - Sir Gangaram Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuaisha M, Itani H, El Masri R, Antoun J. Prevalence of Iron Deficiency (ID) without anemia in the general population presenting to primary care clinics: a cross-sectional study. Postgrad Med. 2020 Apr;132(3):282-287. doi: 10.1080/00325481.2020.1715701. Epub 2020 Jan 22. PMID 31933400
- [Background] Adams J, White M. Characterisation of UK diets according to degree of food processing and associations with socio-demographics and obesity: cross-sectional analysis of UK National Diet and Nutrition Survey (2008-12). Int J Behav Nutr Phys Act. 2015 Dec 18;12:160. doi: 10.1186/s12966-015-0317-y. PMID 26684833
- [Background] Al-Jafar HA. HWA: Hypoferritinemia without anemia a hidden hematology disorder. J Family Med Prim Care. 2017 Jan-Mar;6(1):69-72. doi: 10.4103/2249-4863.214986. PMID 29026752